CLINICAL TRIAL: NCT01324583
Title: An Open Label, Dose Escalation, Safety and Pharmacokinetics Phase I Study With Cabazitaxel Administered as a 1-hour Intravenous Infusion Every 3 Weeks in Combination With Daily Prednisolone in Patients With Hormone Refractory Prostate Cancer
Brief Title: Dose Escalation Study With Cabazitaxel in Combination With Daily Prednisolone in Patients With Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED11576; U1111-1115-4154 (Other: UTN)
Record Dates: First submitted 2011-03-22; First posted 2011-03-29 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabazitaxel; XRP6258; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Patients will receive cabazitaxel as the dose of corresponded level
  1-hour intravenous infusion every 3 weeks plus prednisolone 10 mg orally given daily: Dose Level Cabazitaxel Dose Level -1: 15 mg/m², Level 1: 20 mg/m², Level 2: 25 mg/m²
  Interventions: Drug: Cabazitaxel (XRP6258); Drug: prednisolone

INTERVENTIONS:
Drug: Cabazitaxel (XRP6258) — Pharmaceutical form:solution
  Route of administration: intravenous
Drug: prednisolone — Pharmaceutical form:tablet
  Route of administration: oral

SUMMARY:
Primary Objective:

* To assess the tolerability at global doses

Secondary Objectives:

* Safety
* Pharmacokinetics
* Efficacy

DETAILED DESCRIPTION:
The duration of screening within 28 days, treatment 3 weeks/cycle and follow-up 30 days after the last cabazitaxel administration.

ELIGIBILITY:
Inclusion criteria :

I 01. Diagnosis of histologically or cytologically proven prostate adenocarcinoma, that is refractory to hormone therapy (received prior castration by orchiectomy and/or internal medicine, and documented progression of disease or relapse) who has previously been treated with docetaxel.

I 02. Signed informed consent prior to beginning protocol specific procedures.

I 03. Patients with PSA >20 ng/mL at screening.

Exclusion criteria:

E 01. Age <20 and >74

E 02. ECOG performance status ≥2.

E 03. Prior surgery ≤4 weeks of registration in the study.

E 04. Active secondary cancer including prior malignancy from which the patient has been disease-free for ≤5 years (However, adequately treated superficial basal cell skin cancer before 4 weeks prior to registration can be eligible to the study)

E 05. Inadequate organ function including:

Neutrophils <2.0 x 109/L Platelets <100 x 109/L Hemoglobin <9.0 g/dL (transfusion prohibition within 14 days before registration) Creatinine >1.5 mg/dL. Total bilirubin >1.5 times the upper normal limits of the institutional norms ALT/AST >1.5 times the upper normal limits of the institutional norms

E 06. Previous treatment with <225 mg/m2 cumulative dose of Taxotere® (or docetaxel).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 73 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Identification of maximum tolerated dose | up to 18 months

SECONDARY OUTCOMES:
number of participants with treatment emergent adverse events | up to 18 months
Pharmakokinetic parameters of Cabazitaxel | up to 18 months
Prostate Specific Antigen (PSA) Response | up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (21):
- Japan (21):
  - Investigational Site Number 392011, Bunkyō City
  - Investigational Site Number 392021, Fukuoka
  - Investigational Site Number 392014, Hamamatsu
  - Investigational Site Number 392009, Itabashi-Ku
  - Investigational Site Number 392001, Kashiwa-Shi
  - Investigational Site Number 392020, Kita-Gun
  - Investigational Site Number 392002, Kōtoku
  - Investigational Site Number 392016, Kyoto
  - Investigational Site Number 392017, Kyoto
  - Investigational Site Number 392008, Maebashi
  - Investigational Site Number 392012, Minatoku
  - Investigational Site Number 392015, Nagoya
  - Investigational Site Number 392019, Osaka Sayama-Shi
  - Investigational Site Number 392004, Sapporo
  - Investigational Site Number 392005, Sendai
  - Investigational Site Number 392010, Shinjuku-Ku
  - Investigational Site Number 392018, Suita-Shi
  - Investigational Site Number 392003, Sunto-Gun
  - Investigational Site Number 392007, Tsukuba
  - Investigational Site Number 392006, Yamagata
  - Investigational Site Number 392013, Yokohama

REFERENCES:
- [Derived] Nozawa M, Mukai H, Takahashi S, Uemura H, Kosaka T, Onozawa Y, Miyazaki J, Suzuki K, Okihara K, Arai Y, Kamba T, Kato M, Nakai Y, Furuse H, Kume H, Ide H, Kitamura H, Yokomizo A, Kimura T, Tomita Y, Ohno K, Kakehi Y. Japanese phase I study of cabazitaxel in metastatic castration-resistant prostate cancer. Int J Clin Oncol. 2015 Oct;20(5):1026-34. doi: 10.1007/s10147-015-0820-9. Epub 2015 Mar 26. PMID 25809824